CLINICAL TRIAL: NCT03931707
Title: The China Neonatal Genomes Project
Acronym: CNGP
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: CHFudanU_NNICU11
Record Dates: First submitted 2019-01-28; First posted 2019-04-30 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Newborn; Hereditary Disease; Genetic Predisposition to Disease; Defect, Congenital
Keywords: Newborn; Hereditary Disease; Genetic Predisposition to Disease; Defect, Congenital; Genome Sequencing; Exome Sequencing; Newborn Screening; Genetic Diseases, Inborn
MeSH Terms: conditions — Genetic Diseases, Inborn; Genetic Predisposition to Disease; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Any newborn who joined the newborn genome project, his/her parents will be informed and signed informed consent, in the newborn clinical treatment process to collect venous blood 2ml for gene sequencing and mutation screening.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sick Neonatal Cohort, Sequencing: Infants and their parents enrolled through Neonatal Intensive Care Unit of member hospitals who are un-randomized to receive genomic sequencing. Results disclosure sessions will include a discussion of: family history report, results from standard newborn screening, any potentially medically relevant findings from the baby's medical history/physical exam, and the results of the genomic sequencing report.
  Interventions: Genetic: Genomic sequencing

INTERVENTIONS:
Genetic: Genomic sequencing — Both sick and high-risk newborn un-randomized to receive genomic sequencing will receive a Genomic Newborn Sequencing Report which will include pathogenic or likely pathogenic variants identified in genes associated with childhood-onset disease.

SUMMARY:
The project will carry out the genetic testing of 100000 neonates in the next 5 years. The aim of the project is to construct the Chinese neonatal genome database, establish the genetic testing standard of neonatal genetic diseases, and promote the industrialization of neonatal genetic disease gene testing, improve the training system for genetic counseling.

DETAILED DESCRIPTION:
There are about 900,000 new cases of birth defects in China every year. There are a large number of hereditary diseases, such as primary immune deficiency diseases, genetic metabolic diseases and multiple malformation syndrome, etc. It is important to identify and diagnose these diseases early in life, which can optimize the treatment strategy, improve the quality of life, and achieve the purpose of accurate treatment. To improve the level of diagnosis and prevention of genetic diseases in children is conducive to the birth and education of newborn in our country. The China Neonatal Genome Project is an important part of the China Human single Target Genome Project. The investigators plan to complete genetic testing of 100,000 newborns within 5 years, establish genetic testing standards for genetic diseases of newborns, and promote precise intervention for birth defects. The Genetic Counseling Branch of China Genetics Society, the Pediatrics Hospital affiliated to Fudan University and hundreds of hospitals in China jointly launched the Chinese newborn Genome Project in Shanghai, China. The project will carry out the genetic testing of 100000 neonates in the next 5 years. The study physician and genetic counselor will provide the consultation to families utilizing all available medical information. In the sequencing analysis of the study, this will include the medical history, physical exam, family history, standard newborn screening report. The aim of the project is to construct the Chinese neonatal genome database, establish the genetic testing standard of neonatal genetic diseases, and promote the industrialization of neonatal genetic disease gene testing, improve the training system for genetic counseling.

ELIGIBILITY:
Inclusion Criteria:

* 1. Both parents are of Chinese origin;
* 2. Postnatal age less than 28 days;
* 3. Can be retained to at least 1ml venous blood sample;
* 4. Biological parent or guardian's informed consent.

Exclusion Criteria:

* 1. the nationality of one of the parents is not the Han nationality or other national minorities;
* 2. reluctance of parents to use genetic sequencing data for subsequent research;
* 3. parents under 18 years of age or incapacitated for decision-making;
* 4. subjects older than 28 days.
* 5. multiple pregnancies;
* 6. lack of access to biological samples from which DNA can be extracted;
* 7. failure to sign informed consent

Max Age: 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The subjects were all from all the member organizations participating in the China Newborn Genome Project. They were hospitalized in the neonatal department of each member hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2016-08-08 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of gene sequencing data in neonatal gene bank | From birth to completion of genetic screening, the process last up to 3 months.
  Each newborn that was sequenced was counted as 1. Keep all the data in the gene bank, and finally calculate the number of completed gene sequencing data.
Gene mutation rate | From birth to completion of genetic screening, the process last up to 3 months.
  Taking the number of newborn babies as denominator and the number of neonates with gene mutation detected in gene sequencing as molecules, the whole neonatal gene mutation rate in China was obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhao Zhou, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Dewey FE, Grove ME, Pan C, Goldstein BA, Bernstein JA, Chaib H, Merker JD, Goldfeder RL, Enns GM, David SP, Pakdaman N, Ormond KE, Caleshu C, Kingham K, Klein TE, Whirl-Carrillo M, Sakamoto K, Wheeler MT, Butte AJ, Ford JM, Boxer L, Ioannidis JP, Yeung AC, Altman RB, Assimes TL, Snyder M, Ashley EA, Quertermous T. Clinical interpretation and implications of whole-genome sequencing. JAMA. 2014 Mar 12;311(10):1035-45. doi: 10.1001/jama.2014.1717. PMID 24618965
- [Background] Waisbren SE, Back DK, Liu C, Kalia SS, Ringer SA, Holm IA, Green RC. Parents are interested in newborn genomic testing during the early postpartum period. Genet Med. 2015 Jun;17(6):501-4. doi: 10.1038/gim.2014.139. Epub 2014 Dec 4. PMID 25474344
- [Background] Gilissen C, Hoischen A, Brunner HG, Veltman JA. Unlocking Mendelian disease using exome sequencing. Genome Biol. 2011 Sep 14;12(9):228. doi: 10.1186/gb-2011-12-9-228. PMID 21920049
- [Background] Gonzaga-Jauregui C, Lupski JR, Gibbs RA. Human genome sequencing in health and disease. Annu Rev Med. 2012;63:35-61. doi: 10.1146/annurev-med-051010-162644. PMID 22248320
- [Background] Saunders CJ, Miller NA, Soden SE, Dinwiddie DL, Noll A, Alnadi NA, Andraws N, Patterson ML, Krivohlavek LA, Fellis J, Humphray S, Saffrey P, Kingsbury Z, Weir JC, Betley J, Grocock RJ, Margulies EH, Farrow EG, Artman M, Safina NP, Petrikin JE, Hall KP, Kingsmore SF. Rapid whole-genome sequencing for genetic disease diagnosis in neonatal intensive care units. Sci Transl Med. 2012 Oct 3;4(154):154ra135. doi: 10.1126/scitranslmed.3004041. PMID 23035047
- [Background] Biesecker LG, Green RC. Diagnostic clinical genome and exome sequencing. N Engl J Med. 2014 Sep 18;371(12):1170. doi: 10.1056/NEJMc1408914. No abstract available. PMID 25229935
- [Background] Holm IA, Savage SK, Green RC, Juengst E, McGuire A, Kornetsky S, Brewster SJ, Joffe S, Taylor P. Guidelines for return of research results from pediatric genomic studies: deliberations of the Boston Children's Hospital Gene Partnership Informed Cohort Oversight Board. Genet Med. 2014 Jul;16(7):547-52. doi: 10.1038/gim.2013.190. Epub 2014 Jan 9. PMID 24406460
- [Background] Bhattacharjee A, Sokolsky T, Wyman SK, Reese MG, Puffenberger E, Strauss K, Morton H, Parad RB, Naylor EW. Development of DNA confirmatory and high-risk diagnostic testing for newborns using targeted next-generation DNA sequencing. Genet Med. 2015 May;17(5):337-47. doi: 10.1038/gim.2014.117. Epub 2014 Sep 25. PMID 25255367
- [Derived] Chen X, Chen Y, Xiao T, Dong X, Lu Y, Qian Y, Wang H, Zhou W. CYP2C9*3 Increases the Ibuprofen Response of Hemodynamically Significant Patent Ductus Arteriosus in the Infants with Gestational Age of More Than 30 Weeks. Phenomics. 2021 Nov 11;2(1):72-77. doi: 10.1007/s43657-021-00028-9. eCollection 2022 Feb. PMID 36939774